CLINICAL TRIAL: NCT04775485
Title: FIREFLY-1: A Phase 2, Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of the Oral Pan-RAF Inhibitor DAY101 in Pediatric Patients With RAF-Altered, Recurrent or Progressive Low-Grade Glioma and Advanced Solid Tumors
Brief Title: A Study to Evaluate Tovorafenib in Pediatric and Young Adult Participants With Relapsed or Progressive Low-Grade Glioma and Advance Solid Tumors
Acronym: FIREFLY-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Day One Biopharmaceuticals, Inc. (Industry)
Collaborators: Pacific Pediatric Neuro-Oncology Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAY101-001/PNOC026
Record Dates: First submitted 2021-02-03; First posted 2021-03-01 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Low-grade Glioma; Advanced Solid Tumor
Keywords: Low-grade Glioma; Advanced Solid Tumor; FIREFLY-1; DAY101; Tovorafenib
MeSH Terms: interventions — tovorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Low-Grade Glioma (Experimental): Participants with recurrent or progressive low-grade glioma will receive 420 milligrams/meters square (mg/m^2) of tovorafenib weekly according to dose rounding guidelines and according to their baseline body surface area (BSA).
  Interventions: Drug: Tovorafenib
- Arm 2: Low-Grade Glioma Expanded Access (Experimental): Participants with recurrent or progressive low-grade glioma will receive 420 mg/m^2 of tovorafenib weekly according to dose rounding guidelines and according to their baseline BSA.
  Interventions: Drug: Tovorafenib
- Arm 3: Advanced Solid Tumor (Experimental): Participants with advanced solid tumors will receive 420 mg/m^2) of tovorafenib weekly according to dose rounding guidelines and according to their baseline BSA.
  Interventions: Drug: Tovorafenib

INTERVENTIONS:
Drug: Tovorafenib — Tovorafenib is an oral Type II RAF kinase inhibitor available in 100 mg immediate-release tablet or 25 mg/milliliter (mL) powder for reconstitution.
  Other Names: DAY101

SUMMARY:
This is a Phase 2, multi center, open-label study to evaluate the safety and efficacy of Type II RAF (tovorafenib) in pediatric participants with low-grade glioma or advanced solid tumors. Qualifying genomic alterations will be identified through molecular assays as routinely performed at Clinical Laboratory Improvement Amendments (CLIA) of 1988 or other similarly certified laboratories prior to enrollment into any of the arms. The study will consist of a screening period, a treatment period, a long-term extension phase, end of treatment (EOT) visit(s), a safety follow-up visit, and long-term follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Low Grade Glioma & Low-Grade Glioma Extension: a relapsed or progressive LGG with documented known activating BRAF alteration.
* Advanced Solid Tumor: locally advanced or metastatic solid tumor with documented known or expected to be activating RAF fusion.
* Participants must have histopathologic verification of malignancy at either original diagnosis or relapse.
* Must have received at least one line of prior systemic therapy and have documented evidence of radiographic progression.
* Must have at least 1 measurable lesion as defined by RANO (Arms 1 & 2) or RECIST v1.1 (Arm 3) criteria

Exclusion Criteria:

* Participant's tumor has additional previously-known activating molecular alterations.
* Participant has symptoms of without radiographically recurrent or radiographically progressive disease.
* Known or suspected diagnosis of neurofibromatosis type 1 (NF-1) via genetic testing or current diagnostic criteria.

Other inclusion/exclusion criteria as stipulated by protocol may apply

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 141 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Arm 1: Overall response rate | Up to 48 months
  ORR is defined as percentage of participants with best overall confirmed response of complete response (CR) or partial response (PR) by the Response Assessment in Neuro-Oncology - high-grade glioma (RANO-HGG) criteria.
Arm 2: Number of participants reporting adverse events | Up to 48 months
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Arm 2: Number of participants with clinically significant changes in clinical chemistry parameters | Up to 48 months
Arm 2: Number of participants with clinically significant changes in hematology parameters | Up to 48 months
Arm 3: Overall response rate | Up to 48 months
  Determined by the treating investigator and measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or RANO-HGG criteria, as appropriate.

SECONDARY OUTCOMES:
Arm 1 and 3: Number of participants reporting adverse events | Up to 48 months
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Arm 1 and 3: Number of participants with clinically significant changes in clinical chemistry parameters | Up to 48 months
Arm 1 and 3: Number of participants with clinically significant changes in hematology parameters | Up to 48 months
Arm 1: Area under the concentration-time curve (AUC) of Tovorafenib | Cycle 1: Day 1 and Day 15; Cycles 2, 4, 7, 10 and 13: Day 1
Arm 1: Minimum drug concentration (Cmin) | Cycle 1: Day 1 and Day 15; Cycles 2, 4, 7, 10 and 13: Day 1
Arm 1: Change from Baseline QT interval corrected for heart rate by Fridericia's formula (ΔQTcF) | Baseline to 48 months
Arm 1: Change from Baseline PR interval (ΔPR) | Baseline to 48 months
Arm 1: Change from Baseline QRS interval (ΔQRS) | Baseline to 48 months
Arm 1: Change from baseline heart rate (ΔHR) | Baseline to 48 months
Arm 1: Change in electrocardiogram (ECG) waveform morphology | Baseline to 48 months
Arm 1 and Arm 2: Overall response rate | Up to 48 months
  ORR is defined as percentage of participants with best overall confirmed response of CR or PR by the RANO-HGG criteria.
Arm 1, Arm 2 and Arm 3: Overall response rate in Pediatric participants | Up to 48 months
  ORR is defined as percentage of participants with best overall confirmed response of CR or PR or minor response (MR) by Response Assessment in Pediatric Neuro-Oncology (RAPNO) criteria.CR or PR by RECIST v1.1 criteria.
Arm 1, Arm 2 and Arm 3: duration of progression-free survival (PFS) | Up to 48 months
  PFS as defined by the time following initiation of tovorafenib to progression or death in participants treated with tovorafenib measured by RECIST v1.1, RAPNO, or RANO-HGG criteria as determined by the treating investigator and an IRC.
Arm 1, Arm 2 and Arm 3: Duration of response (DOR) | Up to 48 months
  DOR as defined by the length of response in participants with best overall confirmed response of CR or PR or MR and measured by RANO-HGG, RAPNO, and/or RECIST v1.1 criteria, as applicable.
Arm 1, Arm 2 and Arm 3: Time to response (TTR) | Up to 48 months
  TTR as defined as the time to first response following initiation of tovorafenib in participants with best overall confirmed response of CR or PR measured by RECIST v1.1 or RANO-HGG criteria, as applicable.
Arm 1, Arm 2 and Arm 3: Clinical benefit rate (CBR) | Up to 48 months
  CBR as defined as participants with BOR of CR, PR or stable disease (SD) measured by RECIST v1.1 or RANO-HGG, as applicable, and lasting 12 months or more following initiation of tovorafenib.
Arm 1 and Arm 2: Duration of overall survival | Up to 48 months
  Overall survival as defined by the time following initiation of tovorafenib to death of any cause in participants treated with tovorafenib.
Arm 1: Change from baseline in best corrected visual acuity (BCVA) outcomes | Baseline to 48 months
Arm 1: Changes in molecular analysis of cells obtained from archival tissue | At Screening

CONTACTS AND LOCATIONS:
Locations (35):
- United States (14):
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Doernbecher Children's Hospital Oregon & Health Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (5):
  - Queensland Children's Hospital, Brisbane
  - Royal Children's Hospital, Parkville
  - Perth Children's Hospital, Perth
  - Sydney Children's Hospital, Randwick
  - The Children's Hospital at Westmead, Westmead
- Canada (3):
  - Centre Hospitalier Universitaire Ste-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Mère-Enfant Soleil du CHU, Québec, Quebec
- Rigshospitalet, Copenhagen, Denmark
- Germany (2):
  - Charité Universitätsmedizin Berlin, Campus Virchow Klinikum, Otto-Heubner-Centrum für Kinder, Berlin
  - Hopp-Kindertumorzentrum Heidelberg (KiTZ), KiTZ Clinical Trial Unit (ZIPO), Heidelberg
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
- Princess Maxima Center for Pediatric Oncology, Utrecht, Netherlands
- KK Women's and Children's Hospital, Singapore, Singapore
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital - Yonsei University, Seoul
- Universitäts-Kinderspital Zürich - Eleonorenstiftung, Zurich, Switzerland
- United Kingdom (2):
  - UCL Great Ormond Street Institute of Child Health, London
  - Newcastle University, Newcastle upon Tyne

REFERENCES:
- [Derived] Kilburn LB, Khuong-Quang DA, Hansford JR, Landi D, van der Lugt J, Leary SES, Driever PH, Bailey S, Perreault S, McCowage G, Waanders AJ, Ziegler DS, Witt O, Baxter PA, Kang HJ, Hassall TE, Han JW, Hargrave D, Franson AT, Yalon Oren M, Toledano H, Larouche V, Kline C, Abdelbaki MS, Jabado N, Gottardo NG, Gerber NU, Whipple NS, Segal D, Chi SN, Oren L, Tan EEK, Mueller S, Cornelio I, McLeod L, Zhao X, Walter A, Da Costa D, Manley P, Blackman SC, Packer RJ, Nysom K. The type II RAF inhibitor tovorafenib in relapsed/refractory pediatric low-grade glioma: the phase 2 FIREFLY-1 trial. Nat Med. 2024 Jan;30(1):207-217. doi: 10.1038/s41591-023-02668-y. Epub 2023 Nov 17. PMID 37978284

DOCUMENTS (2):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT04775485/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT04775485/SAP_001.pdf